CLINICAL TRIAL: NCT03670446
Title: Pharmacists' Intervention in Patients Using Novel Oral Anticoagulants：A Study on Behavioral Patterns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018[173]
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Anticoagulants; Intention; Behavioral Symptoms
MeSH Terms: conditions — Behavioral Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacists' intervention (Experimental): A group of participants assigned to a pharmaceutical intervention
  Interventions: Other: Pharmacists' intervention
- Routine therapy (No Intervention): A group of participants assigned to a control (routine therapy)

INTERVENTIONS:
Other: Pharmacists' intervention — 1. Medication education: When the patient is enrolled in the intervention group, pharmacists issue an education manual to give a medical education which contains the reasons for using NOACs, the characteristics of the drug, the precautions, and how to monitor the efficacy. Pharmacists re-educate through telephone or clinic during follow-up.
  2. Establish a medical record and remind their follow-up by message, phone every 2 weeks.
  3. Follow-up in the 4th week and 8th week : Pharmacists recommend patients for drug therapy optimization after conducting a full pharmacotherapy review of each patient's medication regimen and remind them to test urinary occult blood every 1-3 months, detect hemoglobin and liver/kidney function every 3-6 months.
  Arms: Pharmacists' intervention

SUMMARY:
Novel oral anticoagulant drugs (NOACs) are now increasingly used in clinical practice. Although there are outstanding advantages of NOACs, there are also some shortcomings in use. The behavioral pattern of patients using novel oral anticoagulant drugs can directly affect the effect of anticoagulant therapy.

However, at present, there is no study on behavioral patterns of compliance and cognition in patients using NOACs in China. There are few reports on the management outcomes of NOACs anticoagulant therapy as well. Above all, exploring whether pharmacists change behavioral patterns in patients using NOACs is of great significance to improve the effectiveness and safety and to prove the value of pharmacists who provide pharmaceutical care.

DETAILED DESCRIPTION:
The study is a prospective randomized controlled trial. Patients who will use NOACs are prospectively divided into routine group and pharmacist intervention group.

For the intervention group, pharmacists regularly provide telephone and outpatient follow-up combined with patient medication education, establishing database system, telephone reminder, etc. At the 12-week follow-up, behavioral patterns of compliance, self-anxiety, depression status and satisfaction with the pharmacist service will be evaluated in both groups. Pharmacodynamic substitution indicators and endpoints will be collected as well.

Clinical data is designed to be collected from 400 patients, 200 patients each group. Data will be recorded by Epidata dual-track, analyzed by SPSS19.0 software. P<0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients or inpatients with anticoagulation indications of novel oral anticoagulant drugs (NOACs).
2. New prescriptions for NOACs, or previous prescriptions for NOACs, not received any intervention by pharmacists before.
3. Written informed consent was obtained from patients or their families.

Exclusion Criteria:

1. Patients who did not use novel oral anticoagulants.
2. Patients who had received interventions from pharmacists, such as medication education.
3. Written informed consent was not obtained from patients or their families.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 12 weeks
  The Morisky, Green, and Levine Adherence Scale (MGLS) was used to evaluate the medication compliance of dabigatran etexilate and rivaroxaban during treatment. According to the scores of MGLS, compliance was divided into three groups: A score of 0 indicated high compliance; a score of 1 or 2 illustrated intermediate compliance; and a score of 3 or 4 indicated low compliance.
Mental status | 12 weeks
  Mental status is assessed by Self-rating Depression Scale (SDS) and Self-rating Anxiety Scale (SAS).
  The threshold value of depression assessment was 53, the higher the score, the more obvious the tendency of depression. 53-62 is defined as mild depression, 63-72 for moderate depression, 72 points above for severe depression.
  The standard score of SAS was 50, of which 50-59 is mild anxiety, 60-69 is moderate anxiety and 69 is severe anxiety. The patient's awareness of medication is assessed by a self-designed awareness questionnaire.
anti-Xa and IIa activities | 12 weeks
  Anti-Xa/IIa activity test is divided into peak concentration and valley concentration detection; peak concentration is 100 ng/ml as the critical value, Valley concentration is 50 ng/ml as the limit, divided into better or poor pharmacodynamic indicators. patients with peak concentration > 100 ng/ml or valley concentration > 50 ng/ml are defined as better pharmacodynamic indicators.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China Rehabilitation Research Center Beijing Boai Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing